CLINICAL TRIAL: NCT02013024
Title: The Effect of Vitrification Versus Slow Freezing on Day 3: a Randomised Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sophie Debrock (Other)
Responsible Party: Sponsor-Investigator, Sophie Debrock, clinical embryologist PhD, KU Leuven
Organization: KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S53410
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Cryopreservation of Embryos

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- cryopreservation technique (Active Comparator): slow freezing cryopreservation technique
  Interventions: Other: cryopreservation technique
- vitrification cryopreservation technique (Active Comparator): vitrification cryopreservation technique
  Interventions: Other: cryopreservation technique

INTERVENTIONS:
Other: cryopreservation technique

SUMMARY:
Randomized controlled trial (RCT) testing the hypothesis that vitrification is superior to slow freezing.

ELIGIBILITY:
Inclusion Criteria:

* Patients (with female age < 40 years)
* Patients undergoing a 1st oocyte retrieval for an IVF/Intracytoplasmatic Sperm Injection (ICSI) treatment
* Patients planned for an embryo transfer on day 3.
* Patients with supernumerary embryos of sufficient quality for freezing/vitrifying on day 3.
* Fresh personal (own oocytes)
* One inclusion in the study per patient.

Exclusion Criteria:

* Patients undergoing a 2nd or higher ranked oocyte retrieval after a fresh cycle with failed pregnancy.
* Female age ≥ 40 year
* Patients with Preimplantation Genetic Diagnosis (PGD)
* Patients with donor oocytes
* Patients with positive serology whose embryos may not be frozen.
* Patients planned for a transfer on day 2 or day 5.
* Patients receiving assisted hatching in the embryo transfer in the frozen cycles.
* Patients who have been included in the study before.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 417 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Life birth rate per embryo thawed | 3 years

SECONDARY OUTCOMES:
live birth rate per embryo transferred | 3
survival rate | 3 year
implantation rate per embryo transferred | 3 years
implantation rate per embryo thawed | 3 years
abortion rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M D'Hooghe, Prof Dr, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Leuven University Fertility Center, Leuven, Belgium

REFERENCES:
- [Derived] Debrock S, Peeraer K, Fernandez Gallardo E, De Neubourg D, Spiessens C, D'Hooghe TM. Vitrification of cleavage stage day 3 embryos results in higher live birth rates than conventional slow freezing: a RCT. Hum Reprod. 2015 Aug;30(8):1820-30. doi: 10.1093/humrep/dev134. Epub 2015 Jun 18. PMID 26089301